CLINICAL TRIAL: NCT06811792
Title: Intrathecal Therapy for Adult Tuberculous Meningitis: Impact on Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Nie WenJuan, chief physician, Beijing Chest Hospital
Other Study IDs: GCP-TB-2024-9-30
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Tuberculous Meningitis
Keywords: Intrathecal Therapy; Tuberculous Meningitis; Outcome
MeSH Terms: conditions — Tuberculosis, Meningeal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- central nervous system tuberculosis: central nervous system tuberculosis (CNS TB) was confirmed by positive results from traditional microbiological tests or nucleic acid amplification testing for Mycobacterium tuberculosis. Patients without microbiological confirmation were diagnosed based on clinical manifestations. Patients were categorised into two groups based on whether they received standard anti-TB therapy with dexamethasone via spinal canal administration (intrathecal therapy group) or standard anti-TB therapy alone (non-intrathecal therapy group).
  Interventions: Procedure: Intrathecal Therapy

INTERVENTIONS:
Procedure: Intrathecal Therapy — Patients who underwent at least one lumbar puncture and spinal canal administration of glucocorticoids during hospitalisation were classified as receiving intrathecal (IT) therapy. Dexamethasone was the glucocorticoid administered intrathecally at a dose of 5 mg per administration. All patients also received oral or intravenous anti-TB regimens, which included at least isoniazid and rifampicin for drug-sensitive TBM cases. Patients diagnosed with or suspected of having drug-resistant TBM who required second-line anti-TB drugs were excluded from the study.

SUMMARY:
Tuberculous meningitis (TBM) is the most lethal form of tuberculosis (TB). While anti-TB regimens remain the cornerstone of treatment, spinal injection of dexamethasone is considered a potentially effective adjuvant therapy. However, its impact on mortality and disability remains uncertain. This study analysed all TBM patients admitted to Beijing Chest Hospital affiliated with Capital Medical University from January 1, 2010 to December 31, 2023. Patients were categorised into two groups based on whether they received standard anti-TB therapy with dexamethasone via spinal canal administration (intrathecal therapy group) or standard anti-TB therapy alone (non-intrathecal therapy group). Propensity score matching was used to balance baseline characteristics, and one-year mortality and severe disability rates were statistically compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. A positive pathogenic diagnosis of tuberculous meningitis, or clinical diagnosis of tuberculous meningitis, refer to the 《2019 Chinese guidelines for the diagnosis and treatment of central nervous system tuberculosis》; 2. Complete patient information can be found, included patients' demographic characteristics, medical histories, presenting signs and symptoms, clinical course, laboratory test results, diagnostic studies, treatments, complications; 3. Patients can be collected from the time of diagnosis and medication to 12 months.

Exclusion Criteria:

* 1. HIV positive patients (as HIV positive patients in China require diagnosis and treatment in specific healthcare systems); 2. Patients who are unable to collect complete demographic information, diagnostic and treatment information, or treatment outcomes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment Interventions
  Patients who underwent at least one lumbar puncture and spinal canal administration of glucocorticoids during hospitalisation were classified as receiving intrathecal (IT) therapy. Dexamethasone was the glucocorticoid administered intrathecally at a dose of 5 mg per administration. All patients also received oral or intravenous anti-TB regimens, which included at least isoniazid and rifampicin for drug-sensitive TBM cases. Patients diagnosed with or suspected of having drug-resistant TBM who required second-line anti-TB drugs were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 837 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
all-cause mortality within 12 months of treatment initiation | From clear diagnosis to the following 12 months.
  The primary endpoint was all-cause mortality within 12 months of treatment initiation.

SECONDARY OUTCOMES:
Disability rate | 12 months
  The disability rate of tuberculosis meningitis patients within 12 months after diagnosis and treatment.

IPD SHARING:
Plan to Share IPD: No
We have a requirement that hospital information and patient information cannot be shared casually.